CLINICAL TRIAL: NCT06567002
Title: A Study to Evaluate the Pharmacokinetics of Single Dose Formulations of MK-6552 and the Effect of Food in Healthy Study Participants
Brief Title: A Study of MK-6552 and the Effect of Food in Healthy Participants (MK-6552-006)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business Reasons
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 6552-006; MK-6552-006 (Other: MSD)
Record Dates: First submitted 2024-08-20; First posted 2024-08-22 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Sequence 1: (Treatment A) → (Treatment B) → (Treatment C) → (Treatment B) → (Treatment C) (Experimental): Period 1: Participants receive MK-6552 Treatment A single dose administered orally under fasted conditions (Period 1 = 4 days). Period 2: Participants receive MK-6552 Treatment B single dose administered orally under fasted conditions (Period 2 = 4 days). Period 3: Participants receive Treatment C single dose administered orally under fasted conditions (Period 3 = 4 days). Period 4: Participants receive MK-6552 Treatment B single dose administered orally under fed conditions (Period 4 = 4 days). Period 5: Participants receive MK-6552 Treatment C single dose administered orally under fed conditions (Period 5 = 4 days). There will be a minimum 3-day washout between periods.
  Interventions: Drug: MK-6552
- Sequence 2: (Treatment B) → (Treatment C) → (Treatment A) → (Treatment B) → (Treatment C) (Experimental): Period 1: Participants receive MK-6552 Treatment B single dose administered orally under fasted conditions (Period 1 = 4 days). Period 2: Participants receive MK-6552 Treatment C single dose administered orally under fasted conditions (Period 2 = 4 days). Period 3: Participants receive MK-6552 Treatment A single dose administered orally under fasted conditions. (Period 3 = 4 days). Period 4: Participants receive MK-6552 Treatment B single dose administered orally under fed conditions (Period 4 = 4 days). Period 5: Participants receive MK-6552 Treatment C single dose administered orally under fed conditions (Period 5 = 4 days). There will be a minimum 3-day washout between periods.
  Interventions: Drug: MK-6552
- Sequence 3: (Treatment C) → (Treatment A) → (Treatment B) → (Treatment B) → (Treatment C) (Experimental): Period 1: Participants receive MK-6552 Treatment C single dose administered orally under fasted conditions (Period 1 = 4 days). Period 2: Participants receive MK-6552 Treatment A single dose administered orally under fasted conditions. (Period 2 = 4 days). Period 3: Participants receive MK-6552 Treatment B single dose administered orally under fasted conditions (Period 3 = 4 days). Period 4: Participants receive MK-6552 Treatment B single dose administered orally under fed conditions (Period 4 = 4 days). Period 5: Participants receive MK-6552 Treatment C single dose administered orally under fed conditions (Period 5 = 4 days). There will be a minimum 3-day washout between periods.
  Interventions: Drug: MK-6552
- Sequence 4: (Treatment A) → (Treatment C) → (Treatment B) → (Treatment C) → (Treatment B) (Experimental): Period 1: Participants receive MK-6552 Treatment A single dose administered orally under fasted conditions (Period 1 = 4 days). Period 2: Participants receive MK-6552 Treatment C single dose administered orally under fasted conditions (Period 2 = 4 days). Period 3: Participants receive MK-6552 Treatment B single dose administered orally under fasted conditions (Period 3 = 4 days). Period 4: Participants receive MK-6552 Treatment C single dose administered orally under fed conditions (Period 4 = 4 days). Period 5: Participants receive MK-6552 Treatment B single dose administered orally under fed conditions (Period 5 = 4 days). There will be a minimum 3-day washout between periods.
  Interventions: Drug: MK-6552
- Sequence 5: (Treatment B) → (Treatment A) → (Treatment C) → (Treatment C) → (Treatment B) (Experimental): Period 1: Participants receive MK-6552 Treatment B single dose administered orally under fasted conditions (Period 1 = 4 days). Period 2: Participants receive MK-6552 Treatment A single dose administered orally under fasted conditions. (Period 2 = 4 days). Period 3: Participants receive MK-6552 Treatment C single dose administered orally under fasted conditions (Period 3 = 4 days). Period 4: Participants receive MK-6552 Treatment C single dose administered orally under fed conditions (Period 4 = 4 days). Period 5: Participants receive MK-6552 Treatment B single dose administered orally under fed conditions (Period 5 = 4 days). There will be a minimum 3-day washout between periods.
  Interventions: Drug: MK-6552
- Sequence 6: (Treatment C) → (Treatment B) → (Treatment A) → (Treatment C) → (Treatment B) (Experimental): Period 1: Participants receive MK-6552 Treatment C single dose administered orally under fasted conditions (Period 1 = 4 days). Period 2: Participants receive MK-6552 Treatment B single dose administered orally under fasted conditions (Period 2 = 4 days). Period 3: Participants receive MK-6552 Treatment A single dose administered orally under fasted conditions. (Period 3 = 4 days). Period 4: Participants receive MK-6552 Treatment C single dose administered orally under fed conditions (Period 4 = 4 days). Period 5: Participants receive MK-6552 Treatment B single dose administered orally under fed conditions (Period 5 = 4 days). There will be a minimum 3-day washout between periods.
  Interventions: Drug: MK-6552

INTERVENTIONS:
Drug: MK-6552 — Oral Administration

SUMMARY:
The primary purpose of this study is to learn what happens to levels of MK-6552 in the blood when MK-6552 is given in different forms to healthy adult participants under fasted and fed conditions.

ELIGIBILITY:
The main inclusion criteria include but are not limited to the following:

* Be in good health

The main exclusion criteria include but are not limited to the following:

* History of clinically significant endocrine, gastrointestinal (GI), cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases
* History of cancer (malignancy)
* Has received any vaccine starting from 30 days prior to study intervention or is scheduled to receive any vaccine through 30 days following study intervention

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-09-09 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-Time Curve from Time 0 to Last Quantifiable Concentration (AUC0-last) of MK-6552 in a Fasted State | Predose and at designated timepoints approximately up to 3 days postdose
  Blood samples will be collected to determine the AUC0-last of MK-6552.
Area Under the Plasma Concentration-Time Curve from Time 0 to Infinity (AUC0-inf) of MK-6552 in a Fasted State | Predose and at designated timepoints approximately up to 3 days postdose
  Blood samples will be collected to determine the AUC0-inf of MK-6552.
Maximum Concentration (Cmax) of MK-6552 in a Fasted State | Predose and at designated timepoints approximately up to 3 days postdose
  Blood samples will be collected to determine the Cmax of MK-6552.
Concentration at 8 hours (C8h) of MK-6552 in a Fasted State | 8 hours postdose
  Blood samples will be collected to determine the C8h of MK-6552.
Concentration at 16 hours (C16h) of MK-6552 in a Fasted State | 16 hours postdose
  Blood samples will be collected to determine the C16h of MK-6552.
Time to maximum concentration (Tmax) of MK-6552 in a Fasted State | Predose and at designated timepoints approximately up to 3 days postdose
  Blood samples will be collected to determine the Tmax of MK-6552.
Apparent Terminal Half-life (t1/2) of MK-6552 in a Fasted State | Predose and at designated timepoints approximately up to 3 days postdose
  Blood samples will be collected to determine the t1/2 of MK-6552.

SECONDARY OUTCOMES:
AUC0-last of MK-6552 in a Fed or Fasted State | Predose and at designated timepoints approximately up to 3 days postdose
  Blood samples will be collected to determine the AUC0-last of MK-6552.
AUC0-inf of MK-6552 in a Fed or Fasted State | Predose and at designated timepoints approximately up to 3 days postdose
  Blood samples will be collected to determine the AUC0-inf of MK-6552.
Cmax of MK-6552 in a Fed or Fasted State | Predose and at designated timepoints approximately up to 3 days postdose
  Blood samples will be collected to determine the Cmax of MK-6552.
C8h of MK-6552 in a Fed or Fasted State | 8 hours postdose
  Blood samples will be collected to determine the C8h of MK-6552.
C16h of MK-6552 in a Fed or Fasted State | 16 hours postdose
  Blood samples will be collected to determine the C16h of MK-6552.
Tmax of MK-6552 in a Fed or Fasted State | Predose and at designated timepoints approximately up to 3 days postdose
  Blood samples will be collected to determine the Tmax of MK-6552.
t1/2 of MK-6552 in a Fed or Fasted State | Predose and at designated timepoints approximately up to 3 days postdose
  Blood samples will be collected to determine the t1/2 of MK-6552.
Number of participants with one or more adverse events (AE) | Up to approximately day 35
  An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study. The number of participants who experience an AE will be reported.
Number of participants discontinuing from study therapy due to AE | Up to approximately day 35
  An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study. The number of participants who discontinue study treatment due to an AE will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- QPS-MRA, LLC-Early Phase ( Site 0001), South Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com